CLINICAL TRIAL: NCT01113645
Title: The Impact of Cranioplasty on Local and Global Cerebral Blood Flow as Clinical Outcome Prognostic Factor in Patients Undergoing Decompressive Craniectomy for Severe Head Injury.
Brief Title: Impact of Cranioplasty On Cerebral Perfusion
Acronym: CCP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: UC0901; 00006477 (Other: IRB)
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2012-12

CONDITIONS: Head Injuries; Subarachnoid Haemorrhage; Intra-cerebral Haemorrhage; Cerebral Thrombosis; Infarction, Middle Cerebral Artery
Keywords: Decompressive craniectomy; Cranioplasty; Cerebral blood flow; Cerebral hemodynamic; Neurological-cognitive test GOS, FAB, MMSE,; Transcranial Doppler
MeSH Terms: conditions — Craniocerebral Trauma; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Intracranial Thrombosis; Infarction, Middle Cerebral Artery; Fanconi Anemia, Complementation Group B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral perfusion evaluation: All patients are evaluated by GOS (Glasgow Outcome Score) and neurocognitive tests by FAB (frontal assessment battery) and MMSE (mini mental state examination) scores. Hemodynamic monitoring by CT perfusion scan, as well as by trans-cranial Doppler.
  Interventions: Procedure: Cerebral perfusion evaluation

INTERVENTIONS:
Procedure: Cerebral perfusion evaluation — The patient who received a craniectomy is included in the study and an information notice given to him. All patients are evaluated by GOS (Glasgow Outcome Score) and neurocognitive tests by FAB (frontal assessment battery) and MMSE (mini mental state examination) scores 1 week prior and 6 and 24 weeks post cranioplasty. Furthermore, hemodynamic monitoring is performed by CT perfusion scan (with quantitative assessment of global and local cerebral flow) 1 week prior and 6 weeks post cranioplasty, as well as by trans-cranial Doppler 1 week prior and 6 and 24 weeks post cranioplasty.

SUMMARY:
The purpose of this study is to examine the impact of cranioplasty on cerebral hemodynamic and blood flow as prognostic factor in patients receiving decompressive craniectomy for Head injuries, Subarachnoid haemorrhage, intra-cerebral haemorrhage, cerebral dural sinus thrombosis, malignant middle cerebral artery stroke.

DETAILED DESCRIPTION:
Background: The decompressive craniectomy has recently experienced a renewed interest in the international neurosurgical community: the number of patients receiving decompressive craniectomy has remarkably increased over last decades. Nowadays the most widely recognized indications for cranioplasty is aesthetic reconstruction and protection of brain against external injuries; it is usually performed several months after the craniectomy. Unexpected improvements of patients neurological status were noted but this phenomenon remains unexplained. This could be due to the reduction of local cerebral compression caused by atmospheric pressure, to improved cerebrospinal fluid hydrodynamics and possibly to the improvement of local and global cerebral hemodynamics, blood flow and metabolism. Main objective: To evaluate changes in local and global cerebral hemodynamics and blood flow before and after skull bone reconstruction. Patients and Methods: Pilot observational study on 20 patients. Inclusion criteria: Patient over 18 and up to 65 years who underwent decompressive craniectomy after severe head injury, subarachnoid hemorrhage, intracerebral hemorrhage, venous sinus thrombosis with hemorrhage / malignant edema and malignant middle cerebral artery stroke requiring of course reconstructive cranioplasty. Exclusion criteria: Patient not affiliated to the French NHS, pregnant and/or nursing women, patients being allergic to CT scan contrast products. Study Protocol: The patient who received a craniectomy is included in the study and an information notice given to him. All patients are evaluated by GOS (Glasgow Outcome Score) and neurocognitive tests by FAB (frontal assessment battery) and MMSE (mini mental state examination) scores 1 week prior and 6 and 24 weeks post cranioplasty. Furthermore, hemodynamic monitoring is performed by CT perfusion scan (with quantitative assessment of global and local cerebral flow) 1 week prior and 6 weeks post cranioplasty, as well as by trans-cranial Doppler 1 week prior and 6 and 24 weeks post cranioplasty. Expected Benefits: Better knowledge of local and global hemodynamic changes in patients after cranioplasty, its possible impact on neurological outcome and as a prognostic factor. Duration of the inclusion period: 1 year Duration of patient participation: 25 weeks (approximately 6 months) Total duration of the study: 1 year and 25 weeks (about 1 and ½ year) Number of patients: 20 Main endpoints: Evaluation of local and global cerebral hemodynamics and blood flow 6 weeks post cranioplasty by CT perfusion scan and trans-cranial Doppler. Secondary endpoints: - Evaluation of neurological and cognitive performances by GOS, FAB and MMSE scores 1 week prior and 6 and 24 weeks post cranioplasty. - Evaluation of local and global cerebral hemodynamics and blood flow by transcranial Doppler 24 weeks post cranioplasty. Statistical analysis: This is a pilot study whose size was determined on the basis of its feasibility (one year). Besides its own interest, this study will clarify the conditions for a future comparative study comparing different strategies of cranioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age up to 65 years
* Patients receiving a decompressive craniectomy for : severe head injuries, Subarachnoid hemorrhage, intra-cerebral hemorrhage, cerebral dural sinus thrombosis, malignant middle cerebral artery stroke and undergoing to reconstructive cranioplasty
* Patients informed about the study and giving consent

Exclusion Criteria:

* Patients being not assisted by the French NHS
* Patients allergic to CT contrast products
* Pregnant and nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 and up to 65 years who underwent decompressive craniectomy after severe head injury, subarachnoid hemorrhage, intracerebral hemorrhage, venous sinus thrombosis with hemorrhage / malignant edema and malignant middle cerebral artery stroke requiring of course reconstructive cranioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of local and global cerebral hemodynamic and blood flow | at 6 weeks
  1 week prior and 6 weeks post cranioplasty by CT perfusion scan and trans-cranial doppler.

SECONDARY OUTCOMES:
Outcome evaluation by Glasgow Outcome Score (GOS), frontal assessment battery (FAB), and mini mental state examination (MMSE) scores | at 6 and 24 weeks
  at 1 week prior and 6 and 24 weeks post cranioplasty.
Evaluation of local and global cerebral hemodynamic and blood flow | at 24 weeks
  24 weeks post cranioplasty by trans-cranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore CHIBBARO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Neurochirurgie - LARIBOISIERE, Paris, France

REFERENCES:
- [Result] Chibbaro S, Di Rocco F, Mirone G, Fricia M, Makiese O, Di Emidio P, Romano A, Vicaut E, Menichelli A, Reiss A, Mateo J, Payen D, Guichard JP, George B, Bresson D. Decompressive craniectomy and early cranioplasty for the management of severe head injury: a prospective multicenter study on 147 patients. World Neurosurg. 2011 Mar-Apr;75(3-4):558-62. doi: 10.1016/j.wneu.2010.10.020. PMID 21600512